CLINICAL TRIAL: NCT02643225
Title: The Role of Umbilical Cord Thickness, Interventricular Septum Thickness and HbA1C Levels in Prediction of Fetal Macrosomia in Patients With Gestational Diabetes Mellitus
Brief Title: The Role of Umbilical Cord Thickness in Prediction of Fetal Macrosomia in Patients With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Lecturer of Obstetrics and Gynaecology Faculty of Medicine, Ain Shams University, Ain Shams University
Other Study IDs: Diabetes mellitus
Record Dates: First submitted 2015-12-26; First posted 2015-12-31 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pregnant women with gestational diabetes: case group
- non diabetic pregnant women: control group

SUMMARY:
The aim of this work is the prediction of fetal macrosomia by measuring:

1. HbA1C.
2. Umbilical cord thickness.
3. Interventricular septum thickness.

DETAILED DESCRIPTION:
This prospective case control study will be carried out at Ain shams university maternity hospital between April 2015 and October 2015 on 80 patients. The patients will be divided into two groups, 40 pregnant women as case group with gestational diabetes mellitus and 40 non diabetic pregnant women as control group after being approved by the local hospital ethics and research committee. A verbal consent will be taken from each patient.

The following investigation will be performed:

1. Calculation of gestational age will be based on the last reliable menstrual period or ultrasound examination within the first trimester.

   The ultrasound examination will be with Voluson E6 equipped with a 3.5 Hz trans-abdominal probe at fetal medicine unit of maternity hospital Ain Shams University.
2. Ultrasound examination will be performed twice at 27-28 weeks and 36-37 weeks of gestation prospectively.

   During ultrasound, fetal biometry (biparietal diameter, abdominal circumference, femur length) and estimated fetal weight will be calculated automatically according to hadlock's formula additionally, the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device.

   The cross sectional area of Wharton's jelly will be computed by subtracting the cross sectional area of the vessels from that of the umbilical cord and the interventricular septum thickness will be measured.
3. HbA1c levels will be measured for diabetes patients.

All the patients will be subjected to :

1. Full history taking including last menstrual period, medical history and past obstetric history.
2. Detailed general physical history examination and obstetrics examination.
3. Ultrasound examination in fetal medicine unit maternity hospital Ain shams university.
4. Venous blood samples will be taken from patients with gestational diabetes mellitus in clinical pathology department Ain Shams University, to measure the level of HbA1c using immunoassay technique. The patients will be followed up till delivery. The neonates will be weighed and fetal macrosomia will be diagnosed if fetal weight is 4 kg or more.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton gestation.
2. Gestational age over 27 weeks.
3. Intact membranes.
4. Normal umbilical morphology (two arteries and one vein).
5. Diagnosis of gestational diabetes.

Exclusion Criteria:

1. The presence of fetal congenital anomalies.
2. Multifetal pregnancy.
3. Maternal chronic diseases (hypertension, renal disease, cardiac and pulmonary disease, etc.).
4. Patients with a diagnosis such as oligohydramnios , pre-eclampsia and intrauterine growth retardation.
5. Patients who used cigarettes or alcohol during pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective case control study will be carried out at Ain shams university maternity hospital between April 2015 and October 2015 on 80 patients. The patients will be divided into two groups, 40 pregnant women as case group with gestational diabetes mellitus and 40 non diabetic pregnant women as control group after being approved by the local hospital ethics and research committee. A verbal consent will be taken from each patient.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women With Gestational Diabetes: case group
  The investigation will be performed to pregnant women with gestational diabetes
  1. Calculation of gestational age will be based on the last reliable menstrual period or the first trimester ultrasound.
  2. Ultrasound examination will be performed twice at 27-28 weeks and 36-37 weeks of gestation prospectively.
     During ultrasound, fetal biometry (biparietal diameter, abdominal circumference, femur length) and estimated fetal weight will be calculated automatically according to hadlock's formula additionally, the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device.
     The cross sectional area of Wharton's jelly will be computed by subtracting the cross sectional area of the vessels from that of the umbilical cord and the interventricular septum thickness will be measured.
  3. HbA1c levels will be measured for diabetes patients.
- Non Diabetic Pregnant Women: control group
  The investigation will be performed to non diabetic pregnant women:
  1. Calculation of gestational age will be based on the last reliable menstrual period or the first trimester ultrasound.
  2. Ultrasound examination will be performed twice at 27-28 weeks and 36-37 weeks of gestation prospectively.
     During ultrasound, fetal biometry (biparietal diameter, abdominal circumference, femur length) and estimated fetal weight will be calculated automatically according to hadlock's formula additionally, the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device.
     The cross sectional area of Wharton's jelly will be computed by subtracting the cross sectional area of the vessels from that of the umbilical cord and the interventricular septum thickness will be measured.
  3. HbA1c levels will be measured for diabetes patients.
Period: Overall Study
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The patients will be divided into two groups, 40 pregnant women as case group with gestational diabetes mellitus and 40 non diabetic pregnant women as control group after being approved by the local hospital ethics and research committee
Groups:
- Pregnant Women With Gestational Diabetes: case group The investigation will be performed to pregnant women with gestational diabetes
  1. Calculation of gestational age will be based on the last reliable menstrual period or the first trimester ultrasound.
  2. Ultrasound examination will be performed at 36-37 weeks of gestation prospectively.
     During ultrasound, the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device and the interventricular septum thickness will be measured.
  3. HbA1c levels will be measured for participants.
- Non Diabetic Pregnant Women: control group
  The investigation will be performed to non diabetic pregnant women:
  1. Calculation of gestational age will be based on the last reliable menstrual period or the first trimester ultrasound.
  2. Ultrasound examination will be performed at 36-37 weeks of gestation prospectively.
     During ultrasound, the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device and the interventricular septum thickness will be measured.
  3. HbA1c levels will be measured for participants.
- Total: Total of all reporting groups
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7) | 32 (7) | 32 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 40 | 40 | 80
Umbilical Cord Cross-sectional area [Mean (Standard Deviation); unit: cm^2] — the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device at 27-28 weeks of gestation.
  cm^2 | 2.77 (1.19) | 2.06 (.77) | 2.42 (.98)

OUTCOME MEASURES:

1. Secondary Outcome: Umbilical Cordcross-sectional Area
Description: the sonographic cross sectional area of umbilical cord, the umbilical arteries and umbilical vein will be measured in a free loop of the umbilical cord using the software of the ultrasound device.
Time Frame: 36-37 weeks of gestation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women
Number analyzed (Participants) | 40 | 40
cm^2 | 3.03 (1.26) | 2.25 (0.94)

2. Secondary Outcome: Prediction of Fetal Macrosomia by Measuring HbA1C in Participants
Description: Venous blood samples will be taken from participants in clinical pathology department Ain Shams University, to measure the level of HbA1c using immunoassay technique.
Time Frame: 36-37 weeks of gestation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of glycosolated hemoglobin
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women
Number analyzed (Participants) | 40 | 40
percentage of glycosolated hemoglobin | 6.6 (1) | 5.2 (0.5)

3. Secondary Outcome: Interventricular Septum Thickness
Description: The interventricular septum thickness will be measured by ultrasound examination
Time Frame: 36-37 weeks of gestation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women
Number analyzed (Participants) | 40 | 40
mm | 0.85 (0.29) | 0.53 (0.12)

4. Primary Outcome: The Number of Participants Who Were Diagnosed With Fetal Macrosomia (Birth Weight)
Description: The neonates will be weighed and fetal macrosomia will be diagnosed if fetal weight is 4 kg or more.
Time Frame: at birth
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women
Number analyzed (Participants) | 40 | 40
participants | 17 | 0

ADVERSE EVENTS:
Time Frame: from gestational week 27 to birth
Description: Adverse Events were assessed during ultrasound examination
Arm/Group | Pregnant Women With Gestational Diabetes | Non Diabetic Pregnant Women
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No